CLINICAL TRIAL: NCT00739141
Title: A Reduced Intensity Conditioning Regimen and the Transplantation of Unrelated Donor Umbilical Cord Blood in Patients With Hematologic Malignancies.
Brief Title: Conditioning Regimen and the Transplantation of Unrelated Donor Umbilical Cord Blood in Patients With Hematologic Malignancies.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-087
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2021-10

CONDITIONS: Leukemia; Myelodysplastic Syndrome; Non-Hodgkins Lymphoma; Chronic Myelogenous Leukemia; Hodgkins Lymphoma
Keywords: CYCLOPHOSPHAMIDE (CYTOXAN); CYCLOSPORINE A; FLUDARABINE; G-CSF; MYCOPHENOLATE MOFETIL (MMF); THI0TEPA; UMBILICAL CORD BLOOD (UCB); 08-087
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease | interventions — fludarabine; Cyclophosphamide; Thiotepa; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): There are three chemotherapy drugs involved. They are called fludarabine (5 doses), cyclophosphamide (1 dose), and thiotepa (2 doses). Also two days of radiation therapy. This is called Total Body Irradiation or TBI. The TBI if given for two days before, the transplant. On transplant day, the cord blood cells will be given through a catheter. The immune suppressing drugs given are called cyclosporine-A (CSA) and mycophenolate mofetil (MMF). These will be started 3 days before the transplant and will be given through the catheter. Later they can be given as tablets.
  Interventions: Drug: fludarabine, cyclophosphamide, thiotepa, radiation therapy, unrelated donor umbilical cord blood graft

INTERVENTIONS:
Drug: fludarabine, cyclophosphamide, thiotepa, radiation therapy, unrelated donor umbilical cord blood graft — Cyclophosphamide 50 mg/kg/dose x 1 IV day -6 (1 dose) Fludarabine 30 mg/m2/dose x 5 IV days -6 to -2 (5 doses) Thiotepa 5 mg/kg/dose x 2 IV days -5 to -4 (2 doses) TBI 200 cGy/dose x 2 days -2 to -1 (2 doses). On transplant day, the cord blood cells will be given through your catheter. The immune suppressing drugs you will receive are called cyclosporine-A (CSA) and mycophenolate mofetil (MMF). These will be started 3 days before the transplant and will be given through your catheter. Later they can be given as tablets.

SUMMARY:
The traditional way of doing a donor transplant is to give high doses of chemotherapy and radiation before giving the stem cells. However, high doses of chemotherapy and radiation can have serious side-effects. The doctors think that the transplant will be safer and more likely to be successful with reduced doses of chemotherapy and radiation. The purpose of this study is to find out how good a combination of chemotherapy and radiation at reduced doses followed by a cord blood transplant are at treating cancer.

The stem cells chosen for the transplant are from umbilical cord blood. Umbilical cord blood is collected from healthy newborn babies and frozen. One cord blood collection is called a "cord blood unit." On transplant day, the cord blood will be given through the catheter just like a blood transfusion. Transplants done this way have been successful. However, this type of transplant is fairly new. Therefore, it is important to study it so the doctors can better understand how it works.

Most blood or bone marrow transplants using donor stem cells are done as part of a study. When patients are on a study we test new ways of treating them which we think may be better than the old ways. We collect information about the result of this treatment so we can understand how well the treatment works. This is so we can learn better ways to treat our patients.

ELIGIBILITY:
Inclusion Criteria:

* At least one cycle of induction or re-induction chemotherapy or lymphoma chemotherapy or azacitidine or decitabine or tyrosine kinase inhibitor.
* Patients aged 18-70 years at initial referral with no available and suitably matched related or unrelated donor.
* Acute myelogenous leukemia (AML):
* Complete first remission (CR1) at high risk for relapse such as:
* Known prior diagnosis of myelodysplasia (MDS) or myeloproliferative disorder;
* Therapy related AML;
* White cell count at presentation > 100,000;
* Presence of extramedullary leukemia at diagnosis;
* Any unfavorable sub type by FAB or WHO classification;
* High-risk cytogenetics (eg those associated with MDS, abnormalities of 5, 7, 8, Philadelphia chromosome, complex karyotype)or high risk molecular abnormalities;
* Requirement for 2 or more inductions to achieve CR1.
* Any patient with newly diagnosed AML with intermediate risk cytogenetics.
* Any patient unable to tolerate consolidation chemotherapy as would have been deemed appropriate by the treating physician.
* Complete second remission (CR2).
* Other acute leukemias that are ambiguous lineage or of other types eg blastic plasmacytoid dendritic cell neoplasm in CR1 or CR2
* Acute lymphoblastic leukemia (ALL):
* lymphoblastic leukemia (ALL):
* Complete first remission (CR1) at high risk for relapse such as:
* White cell count at presentation > 30,000 for B-cell lineage and >100,000 for Tcell lineage;
* Presence of a high-risk cytogenetic abnormality such as t(9;22), t(1;19), t(4;11) or other MLL rearrangements (11q23)or other high-risk molecular abnormality;
* Failure to achieve complete remission after four weeks of induction therapy;
* Any patient with newly diagnosed ALL > or = to 50 years-old;
* Any patient unable to tolerate consolidation and/or maintenance chemotherapy as would have been deemed appropriate by the treating physician.
* Complete second remission (CR2).
* Myelodysplastic Syndrome (MDS):
* Intermediate-1 International Prognostic Scoring System (IPSS) score with poor risk cytogenetics as defined by IPSS.
* Intermediate- 2 or High International Prognostic Scoring System (IPSS) score.
* MDS/ myeloproliferative disorder overlap syndromes.
* Any score with life threatening cytopenia(s), including red cell or platelet transfusion dependence.
* Receipt of at least one cycle of cytotoxic chemotherapy, azacitidine or decitabine.
* MDS patients must have < or = to 5% bone marrow myeloblasts and ANC > or = to 0.2 (growth factor supported if necessary) at transplant work-up.
* Myeloproliferative Disorder (MPD)
* Life-threatening cytopenia(s), and/or red blood cell or platelet transfusion dependence
* Patients with aplasia
* Patients with excess blasts less than or equal to 10% blasts in the bone marrow at work-up.
* Chronic myelogenous leukemia (CML) patients who have failed or are intolerant of tyrosine kinase inhibitors or patients with other myeloproliferative diseases who are high risk and the intent of therapy is cure.
* Any Non-Hodgkins lymphoma (including chronic lymphocytic leukemia)or Hodgkin's lymphoma at high-risk of relapse
* Eligible patients with DLC NHL will:

have relapsed disease following initial therapy but failed to mobilize or had bone marrow involvement and therefore are not suitable for an autologous transplant OR

* have failed an autologous transplant and be in CR after salvage chemotherapy.
* Eligible patients with transformed indolent NHL/CLL will:

have CR/PR of the large cell component of their disease after either salvage chemotherapy or an autologous transplant.

* Eligible patients with mantle cell NHL will:

be high-risk as such as p53 positivity and be in 1st CR/PR after initial therapy OR have relapsed disease following initial therapy and be in 2nd or 3rd CR/PR after salvage chemotherapy.

* Eligible patients with indolent B cell NHL (such as, but not limited to, follicular, small cell or marginal zone NHL) or CLL will have 2nd or subsequent progression (pre-allograft cytoreduction necessary but CR/PR not required).
* Eligible patients with HL will be without progression of disease (POD) after salvage chemotherapy.
* Timing of UCBT:
* Admission for UCBT must be within an acceptable time period after the pre-allograft chemotherapy.
* Organ Function and Performance Status Criteria:
* Karnofsky score > or = to 70 %.
* calculated creatinine clearance > or = to 60 ml/min
* bilirubin < than or = to 1.5 mg/dL, ALT < than or = to 3 x upper limit of normal unless benign congenital hyperbilirubinemia,
* pulmonary function (spirometry and corrected DLCO) > or = to 50% predicted.
* left ventricular ejection fraction > or = to 50%.
* albumin > or = to 3.0.
* Graft Criteria:
* 2 UCB units selected according to current MSKCC unit selection algorithm. High resolution 8 allele HLA typing will be performed. Unit selection will occur based on 8 allele HLA-match and CD34+ dose.
* In addition, each unit will have a cryopreserved dose of at least 1.5 x 10^7 total nucleated cells/recipient body weight (TNC/kg).
* Units with attached segments for confirmatory typing will be given preference.

Exclusion Criteria:

* Diagnosis: acute leukemia in morphologic relapse or with morphologic persistent disease (cytogenetic or molecular persistence/relapse in morphologic CR are eligible); MDS or CML or other myeloproliferative disorder with > 5% blasts; Aggressive lymphoma or HL with POD after salvage chemotherapy.
* Two prior stem cell transplants of any kind.
* One prior autologous stem cell transplant within the preceding 12 months.
* One prior allogeneic stem cell transplant within the preceding 24 months.
* Prior radiation therapy with 400cGy or more of TBI.
* Active and uncontrolled infection at time of transplantation.
* HIV infection.
* Seropositivity for HTLV-1.
* Inadequate performance status/ organ function.
* Pregnancy or breast feeding.
* Patient or guardian unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up, and research tests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-08-12 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Barker, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Ponce DM, Sauter C, Devlin S, Lubin M, Gonzales AM, Kernan NA, Scaradavou A, Giralt S, Goldberg JD, Koehne G, Perales MA, Young JW, Castro-Malaspina H, Jakubowski A, Papadopoulos EB, Barker JN. A novel reduced-intensity conditioning regimen induces a high incidence of sustained donor-derived neutrophil and platelet engraftment after double-unit cord blood transplantation. Biol Blood Marrow Transplant. 2013 May;19(5):799-803. doi: 10.1016/j.bbmt.2013.02.007. Epub 2013 Feb 14. PMID 23416850
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Hematologic Malignancies: There are three chemotherapy drugs involved. They are called fludarabine (5 doses), cyclophosphamide (1 dose), and thiotepa (2 doses). Also two days of radiation therapy. This is called Total Body Irradiation or TBI. The TBI if given for two days before, the transplant. On transplant day, the cord blood cells will be given through a catheter. The immune suppressing drugs given are called cyclosporine-A (CSA) and mycophenolate mofetil (MMF). These will be started 3 days before the transplant and will be given through the catheter. Later they can be given as tablets.
Period: Overall Study
Arm/Group | Participants With Hematologic Malignancies
Started | 86
Completed | 81
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Hematologic Malignancies
Number analyzed (Participants) | 86
Age, Continuous [Median (Full Range); unit: years] | 51 [25 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 80
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 53
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival/PFS at 1 Year Post UCBT.
Description: To obtain a preliminary estimate of progression free survival at 1 year post UCBT. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1 year post UCBT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With Hematologic Malignancies
Number analyzed (Participants) | 86
percentage of participants | 84 [77 to 92]

2. Secondary Outcome: Number of Participants With Neutrophil Recovery Post Allograft for Haplo-dCBT Recipients
Description: Successful primary donor engraftment = neutrophill recovery within the first 45 days after transplant and partial/complete donor chimerism (>/= 10%)
Time Frame: up to 13 days from engraftment
Population: 43 haplo-dCBT recipients in this analysis 43 dCBT recipient
Measure: Number; unit: participants
Arm/Group | Participants With Hematologic Malignancies
Number analyzed (Participants) | 86
participants
  Haplo-dCBT with early haplo-derived myeloid bridge | 17
  Haplo-dCBT with transient haplo-derived bridge with second neutrophil nadir | 13
  Haplo-dCBT with no bridge | 13
  Remaining dCBT recipient | 43

3. Secondary Outcome: Percentage of Participants With Sustained CB-derived Neutrophil Engraftment
Description: The day 100 cumulative incidence of sustained CB-derived neutrophil engraftment.
Time Frame: 100 days
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With Hematologic Malignancies
Number analyzed (Participants) | 86
Percentage of participants | 99 [87 to 99]

4. Secondary Outcome: Percentage of Participants With Sustained CB-derived Platelet Engraftment
Description: The day 100 cumulative incidence of sustained CB-derived platelet engraftment to >/= 20 x 10^9/L
Time Frame: 100 days
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With Hematologic Malignancies
Number analyzed (Participants) | 86
Percentage of participants | 93 [85 to 97]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Participants With Hematologic Malignancies
All-Cause Mortality (participants affected / at risk) | 36/86
Serious Adverse Events (participants affected / at risk) | 41/86
Other Adverse Events (participants affected / at risk) | 47/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Hematologic Malignancies (N=86)
Anorexia (Metabolism and nutrition disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Blood/Bone Marrow, other (Blood and lymphatic system disorders) | 1
Creatinine (Investigations) | 1
Death not assoc w CTCAE term- Death NOS (General disorders) | 26
Death not assoc w CTCAE term- Multi-organ failure (General disorders) | 3
Death not assoc w CTCAE term- Sudden death (General disorders) | 1
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 4
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1
Fever (in the absence of neutropenia) (General disorders) | 2
Gastrointestinal, other (Gastrointestinal disorders) | 1
Hemoglobin (Investigations) | 1
Hemolysis (Blood and lymphatic system disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Infection w/ Gr 3/4 neut, Blood (Infections and infestations) | 1
Infection, other (Infections and infestations) | 10
Muscle weakness - Whole body/general (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Neurology - Other (specify) (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - Cardiac/heart (Cardiac disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Pain - Urethra (Renal and urinary disorders) | 1
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Renal/Genitourinary-Other Specify (Renal and urinary disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Weight loss (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Hematologic Malignancies (N=86)
ALT, SGPT (Investigations) | 20
AST, SGOT (Investigations) | 9
Alkaline phosphatase (Investigations) | 6
Bilirubin (hyperbilirubinemia) (Investigations) | 37
Creatinine (Investigations) | 7
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 47
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT00739141/Prot_SAP_000.pdf